CLINICAL TRIAL: NCT01150526
Title: Efficacy of a New Delivery System for Beta-hydroxy-beta-methylbutyrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MTI2010-CS02
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Acute Exercise; Muscle Inflammation; CaHMB; HMB Free Acid Gel; Healthy Subjects
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Oral Placebo capsule and one placebo gel dosage given 30 min prior to the acute exercise session. A placebo capsule and placebo gel dosage are then administered 3 times daily during the remainder of the study.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Placebo Gel Dosage
- CaHMB Pre (Experimental): Oral CaHMB capsule and one placebo gel dosage given 30 min prior to the acute exercise session. A placebo capsule and placebo gel dosage are then administered 3 times daily during the remainder of the study.
  Interventions: Dietary Supplement: CaHMB; Dietary Supplement: Placebo; Dietary Supplement: Placebo Gel Dosage
- CaHMB Pre and Post (Experimental): Oral CaHMB capsule and one placebo gel dosage given 30 min prior to the acute exercise session. A CaHMB capsule and placebo gel dosage are are then administered 3 times daily during the remainder of the study.
  Interventions: Dietary Supplement: CaHMB; Dietary Supplement: Placebo Gel Dosage
- HMB Free Acid Gel Pre (Experimental): Oral placebo capsule and one HMB free acid gel dosage given 30 min prior to the acute exercise session. A placebo capsule and placebo gel dosage are then administered 3 times daily during the remainder of the study.
  Interventions: Dietary Supplement: HMB Free Acid Gel; Dietary Supplement: Placebo; Dietary Supplement: Placebo Gel Dosage
- HMB Free Acid Gel Pre and Post (Experimental): Oral placebo capsule and one HMB free acid gel dosage given 30 min prior to the acute exercise session. A placebo capsule and HMB free acid gel dosage are then administered 3 times daily during the remainder of the study.
  Interventions: Dietary Supplement: HMB Free Acid Gel; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CaHMB — CaHMB capsules with each capsule containing 0.8 g of HMB
  Arms: CaHMB Pre; CaHMB Pre and Post
Dietary Supplement: HMB Free Acid Gel — HMB Free acid in a gel form with each dose supplying 0.8 g of HMB free acid
  Arms: HMB Free Acid Gel Pre; HMB Free Acid Gel Pre and Post
Dietary Supplement: Placebo — Placebo capsules similar in size and color to the CaHMB capsules used in the study
  Arms: CaHMB Pre; HMB Free Acid Gel Pre; HMB Free Acid Gel Pre and Post; Placebo
Dietary Supplement: Placebo Gel Dosage — A corn syrup based placebo with flavoring and taste similar to the HMB Free Acid Gel
  Arms: CaHMB Pre; CaHMB Pre and Post; HMB Free Acid Gel Pre; Placebo

SUMMARY:
The proposed study will test efficacy of HMB in free acid gel to decrease muscle damage, diminish inflammatory response, and improve muscle strength recovery following an acute exercise stress. HMB in a free acid gel or in CaHMB capsule form will be administered as either a single dose before a bout of acute exercise or in multiple doses (one before and three daily doses for the 4 days following the acute exercise). We hypothesize that HMB in free acid gel will result in less muscle damage, diminished inflammatory response, and improved muscle strength recovery than either a placebo or CaHMB treatment following a bout of acute eccentric exercise. Our endpoints will include measurements of: (1) markers for muscle damage (CPK and LDH); (2) indicators of inflammation (CRP, TNF-α, IL-6, IL-1ra and IL-18); and (3) muscle strength recovery and soreness.

ELIGIBILITY:
Inclusion Criteria:

* Must live within 50 miles of Ames, Iowa
* Free of cardiac, liver, pulmonary, and kidney disease
* Free of chronic inflammatory disease including rheumatoid arthritis, osteoarthritis, inflammatory bowel disease, and psoriasis
* Free diabetes mellitus
* Not classified as morbidly obese (BMI must be less than 40)
* Free of cardiac, liver, pulmonary, and kidney disease
* No other serious medical illness
* Normal menstrual cycle and not pregnant or lactating
* Able to consume supplements and perform required exercise testing

Exclusion Criteria:

* Live more than 50 miles from Ames, Iowa
* Presence of cardiac, liver, pulmonary, and kidney disease
* Presence of chronic inflammatory disease including rheumatoid arthritis, osteoarthritis, inflammatory bowel disease, and psoriasis
* Diabetes mellitus
* Classified as morbidly obese (BMI is greater than 40)
* No other serious medical illness
* Abnormal menstrual cycle, pregnant or lactating
* Not able to consume supplements and perform required exercise testing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Decrease in muscle damage and inflammation | 4 days post eccentric exercise bout
  Serum analysis for markers of muscle damage (CPK) and inflammation (IL-6, IL-18, IL1ra, TNF-a, CRP) will be measured at 24, 48, 72, and 96 h post exercise bout

SECONDARY OUTCOMES:
Improvement in strength recovery and decrease in soreness | 4 days post eccentric exercise bout
  Muscle strength recovery and soreness will be measured at 24, 48, 72, and 96 h post exercise bout.

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Iowa State University, Ames, Iowa, United States